CLINICAL TRIAL: NCT00542087
Title: A Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Etoricoxib 60 mg and Diclofenac Sodium 150 mg in Patient With Osteoarthritis of the Knee or Hip
Brief Title: Etoricoxib vs. Diclofenac in OA (0663-805)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-805; 2007_625; NCT00092794 (obsolete NCT alias)
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib / Duration of Treatment: 6 Weeks
Drug: Comparator: diclofenac sodium / Duration of Treatment: 6 Weeks

SUMMARY:
To compare the safety and tolerability of etoricoxib and diclofenac sodium in the treatment of osteoarthritis of the knee or hip during a six week period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 40 years old and diagnosed with osteoarthritis of the knee or hip
* Has a history of treatment with NSAIDs with positive therapeutic benefit
* Agree to limit alcohol intake to less than 7 drinks per week and avoid unusual strenuous activity
* Females who are able to have children must have negative urine pregnancy tests

Exclusion Criteria:

* Has rheumatoid arthritis, lupus, Paget's disease affecting the study joint, or Wilson's disease
* History of acute ligament or meniscus damage to the study joint (knee or hip) within the past 2 years or arthroscopic surgery on the affected study joint with the past 6 months
* Requires joint replacement

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2002-03-22 (Actual); Primary Completion 2002-12-20 (Actual); Study Completion 2002-12-20 (Actual)

PRIMARY OUTCOMES:
This study will assess the effectiveness of the study drug vs. a comparator to treat successfully OA-related joint pain (judged by WOMAC pain subscale).

SECONDARY OUTCOMES:
The study drug will be safe and well tolerated during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Zacher J, Feldman D, Gerli R, Scott D, Hou SM, Uebelhart D, Rodger IW, Ozturk ZE; etoricoxib OA study group. A comparison of the therapeutic efficacy and tolerability of etoricoxib and diclofenac in patients with osteoarthritis. Curr Med Res Opin. 2003;19(8):725-36. doi: 10.1185/030079903125002469. PMID 14687444